CLINICAL TRIAL: NCT05518279
Title: Early Administration Of Tranexamic Acid And Acute Blood Loss In Patients With Hip Fractures: A Prospective, Randomized, Double-blinded, Placebo Controlled Trial
Brief Title: Early Administration Of Tranexamic Acid And Acute Blood Loss In Patients With Hip Fractures
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Could not work out internal logistics
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Trent Guthrie, Department of Orthopaedic Surgery, Trauma Division; Program Director: Orthopaedic Surgery Residency, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11411
Record Dates: First submitted 2019-01-22; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Hip Fractures; Blood Loss
Keywords: hip fracture; blood loss; tranexamic acid
MeSH Terms: conditions — Hip Fractures; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both participants and treatment team will be blinded to the treatment medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic Acid Treatment Group (Active Comparator): The intervention for the treatment group is as follows: participants in this treatment arm will given 1950mg of oral tranexamic acid pills (3 tablets, 650mg each) in the emergency department following diagnosis of hip fracture.
  Interventions: Drug: Tranexamic Acid Pill
- Oral Placebo Control Group (Placebo Comparator): The intervention for the control group is as follows: participants in this treatment arm will given 3 tablets of oral placebo pills in the emergency department following diagnosis of hip fracture.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tranexamic Acid Pill — Patients will receive 1950mg of an oral tranexamic acid pill (3 pills total) while down in the Emergency Department after being diagnosed with a hip fracture. After they receive the oral TXA and are medically optimized, they will be taken to the operating room for fracture fixation.
  Arms: Tranexamic Acid Treatment Group
Drug: Placebo Oral Tablet — Patients in the control arm will receive 3 placebo pills while down in the Emergency Department after being diagnosed with a hip fracture. After they receive the placebo pills and are medically optimized for surgery, they will be taken to the operating room for fracture fixation.
  Arms: Oral Placebo Control Group

SUMMARY:
The study is a prospective, randomized, double blinded, placebo controlled trial that aims to investigate the hypothesis that early administration of tranexamic acid (TXA) following diagnosis of hip fracture will lower pre and postoperative blood loss and transfusion rates. Patients who present to the hospital with a hip fracture will be recruited and randomized into two treatment arms. The treatment group will receive 1950mg of oral TXA (three tablets, 650 mg each) and the control group will be given three tablets of oral placebo while in the Emergency Department. Patients will then be admitted to the Orthopaedic Trauma service and treated surgically with cephalomedullary nail, hemiarthroplasty, sliding hip screw, percutaneous screws, or total hip arthroplasty.

DETAILED DESCRIPTION:
There remains a high incidence of blood transfusion in patients following hip fractures. Tranexamic acid (TXA) has well-studied efficacy in decreasing blood loss and transfusion requirements in the context of general trauma, as well as several elective orthopaedic procedures. Although blood is lost in hip fracture surgery itself, it is also known that there is significant blood loss pre-operatively following the hip fracture event, particularly in extracapsular hip fractures. A prospective, randomized, double blinded, placebo controlled trial will elucidate the roll of early administration of TXA in a population of patients who sustain hip fractures. The study aims to investigate the hypothesis that early administration of TXA following diagnosis of hip fracture will lower pre and postoperative blood loss and transfusion rates. There will be two treatment arms in the study. The treatment group will be given 1950mg of oral TXA (3 tablets, 650mg each) in the emergency department following diagnosis of hip fracture. Those randomized to the control group will be given 3 tablets of oral placebo in the emergency department following diagnosis of hip fracture. Patients will then be admitted to the Orthopaedic Trauma service and treated surgically with cephalomedullary nail, hemiarthroplasty, sliding hip screw, percutaneous screws, or total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50
* Clinical diagnosis of acute femoral neck, intertrochanteric or subtrochanteric femur fracture

Exclusion Criteria:

* anticoagulant use at time of admission to emergency department
* documented allergy to tranexamic acid
* history of deep vein thrombosis or pulmonary embolism
* hepatic dysfunction (aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 60)
* renal dysfunction (Creatinine > 1.5 or Glomerular Filtration Rate < 30)
* active coronary artery disease (event within 12 months)
* history of cerebral vascular accident within 12 months
* presence of drug eluting stent
* color blindness
* active cancer
* coagulopathy (International Normalized Ratio > 1.4, Partial Thromboplastin Time > 1.4 times normal, platelets < 50,000)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Blood transfusion rate | This outcome will be recorded daily from the time of admission to the Emergency Department through the time of discharge from the hospital, assessed up to 7 days.
  Preoperative, intraoperative, and postoperative blood transfusions will be considered as the primary outcome measure. This outcome will be measured in number of units of packed red blood cells administered during the participant's hospital stay.
Hemoglobin Level | This outcome will be recorded daily from the time of admission to the Emergency Department to the time of discharge from the hospital, up to 7 days.
  Labs, specifically a complete blood count (CBC) to evaluate a hemoglobin level (in grams per deciliter), will be drawn at the following time points: Admission to the Emergency Department, nightly (9pm) for each day of hospitalization and one hour after completion of a blood transfusion.

SECONDARY OUTCOMES:
Estimated blood loss | Starting at time of surgical incision and will end once the surgery is completed.
  Measured amount of blood loss recorded during the surgery. These values will be compared between the two study arms to determine if administration of oral TXA decreases the intra-operative blood loss.
Frequency of adverse events. | From time of admission to the Emergency department up to 12 months after the date of surgery. Outcome measure will be recorded daily while participant is hospitalized and monthly after discharge from the hospital.
  Documentation of any adverse events in the peri-operative period. For example, transfusion reaction, myocardial infarction, symptomatic deep vein thrombosis, pulmonary embolism, stroke, reoperation, readmission, infection, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Trent Guthrie, MD, Principal Investigator — Henry Ford Hospital Department of Orthopaedic Surgery

IPD SHARING:
Plan to Share IPD: No